CLINICAL TRIAL: NCT04720573
Title: Influence of the Neuromuscular Blockade and Its Reversal on Perioperative Arrhythmias
Brief Title: Reversal of Neuromuscular Blockade and Perioperative Arrhythmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: Medipol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BasaksehirCamSakuraSehirH
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Neuromuscular Blockade
Keywords: Bradycardia; Cardiac Arrhythmias; Neostigmine; Neuromuscular Blockade; Sugammadex; Train-of-Four Monitoring
MeSH Terms: conditions — Bradycardia; Arrhythmias, Cardiac | interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Investigator
Masking Description: The investigator assessing the ECGs, and rhythm holter recordings was blinded to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group N (Active Comparator): Neostigmine was used for the reversal of neuromuscular blockade.
  Interventions: Drug: Neostigmine
- Group S (Active Comparator): Sugammadex was used for the reversal of neuromuscular blockade.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine — 50 mcg/kg neostigmine was used under the guidance of TOF monitoring after cessation of anesthesia.
  Arms: Group N
Drug: Sugammadex — 2 mg/kg sugammadex was used under the guidance of TOF monitoring after cessation of anesthesia.
  Arms: Group S

SUMMARY:
Patients scheduled for elective abdominopelvic laparoscopic surgery under general anesthesia were included. Rocuronium was used for the neuromuscular blockade (NMB) and the level of NMB was monitored with train-of-four (TOF) measurements. The participants from whom informed consent had been received were allocated to two groups according to the agent used for reversal of NMB, sugammadex, or neostigmine. The ECG recordings of the subjects were followed with a rhythm Holter device throughout the procedure until the postoperative 12th hour. Additionally, preoperative and immediate postoperative 12-lead ECGs were evaluated for corrected QT calculations and QT dispersion. Proarrhythmogenicity was assessed with QT related measurements. The documented arrhythmic events on the Holter monitoring were designated as clinical end-points.

DETAILED DESCRIPTION:
Eighty consecutive patients, to whom an elective abdominopelvic surgery under general anesthesia was planned, were included in the study. Participants were allocated to two groups considering the agent to be used for the reversal of neuromuscular blockade by closed-envelope randomization. Neostigmine was used for this purpose in Group N, while sugammadex was used in Group S. Demographic features including hypertension, diabetes mellitus, presence of coronary artery disease, heart failure, and previous arrhythmia were noted. Body mass index was calculated with the Du Bois method. In the operation room, heart rate, blood pressure, body temperature, arterial oxygen saturation, and TOF ratio were recorded. General anesthesia was induced with midazolam, fentanyl, and propofol; and maintained by remifentanil and sevoflurane. In Group N, 50 mcg/kg neostigmine and 20 mcg/kg atropine were used for NMB reversal. In Group S, reversal was achieved by the administration of sugammadex at a dose of 2 mg/kg. QT interval was measured in leads DII or V5 and adjusted to the heart rate by the Bazzett formula. QTc values at the baseline and postoperative ECGs were recorded and presented with milliseconds. An increase of over 60 ms in QTc interval or a postoperative measurement over 500 ms were assumed to be distinctly abnormal. QT dispersion was calculated by extracting the minimum QT length from the maximum QT length in 12-lead ECG. In rhythm holter monitoring, minimum and mean heart rates and specific arrhythmic events were recorded. In the heart rate variability analysis, the standard deviation of the interbeat intervals of normal sinus beats (SDNN) and the root mean square of successive differences between normal heartbeats (rMSSD) were calculated. The following events were designated as clinical end-points.

* Pause (no waves on ECG recording at least for 3 seconds)
* Significant bradycardia (sinus bradycardia persisted at least for 30 seconds with a rate below 50 beats/min)
* High-grade atrioventricular block (2nd-degree Mobitz Type II or 3rd degree)
* Supraventricular tachycardia (sudden onset tachycardia with narrow QRS complexes persisted over 30 seconds)
* Atrial flutter or fibrillation (sustained over 30 seconds)
* Frequent premature ventricular beats (≥30 beats/hour)
* Any ventricular tachycardia (wide QRS complexes)

ELIGIBILITY:
Inclusion Criteria:

* Planned abdominopelvic surgery under general anesthesia
* ASA II-IV
* Willing to give consent

Exclusion Criteria:

* Significantly impaired left ventricular systolic function (ejection fraction < 40%)
* Significant ongoing arrhythmia (sinus bradycardia with a heart rate below 40 beats/min, Mobitz Type II or 3rd-grade atrioventricular block, persistent or permanent atrial flutter or fibrillation, bigeminal or trigeminal ventricular premature beats, documented ventricular tachycardia)
* Severely reduced renal function (glomerular filtration rate < 30 ml/min/1.73 m2)
* Severe respiratory diseases, neuromuscular disorders, and known allergy to anesthetic agents or adjuvants
* Pregnancy and breastfeeding
* Observing the typical signs of a channelopathy (short QT syndrome, long QT syndrome, Brugada syndrome, etc.) and history of recent medical therapy with agents exhibiting a high probability of QT prolongation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Significant arrhythmic event | Up to 12 hours after surgical procedure
  Pause (no waves on ECG recording at least for 3 seconds), significant bradycardia (sinus bradycardia persisted at least for 30 seconds with a rate below 50 beats/min), high-grade atrioventricular block (2nd-degree Mobitz Type II or 3rd degree), supraventricular tachycardia (sudden onset tachycardia with narrow QRS complexes persisted over 30 seconds), atrial flutter or fibrillation (sustained over 30 seconds), Frequent premature ventricular beats (≥30 beats/hour).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorentz MN, Vianna BS. Cardiac dysrhythmias and anesthesia. Rev Bras Anestesiol. 2011 Nov-Dec;61(6):798-813. doi: 10.1016/S0034-7094(11)70090-3. English, Multiple languages. PMID 22063382
- [Background] Dahl V, Pendeville PE, Hollmann MW, Heier T, Abels EA, Blobner M. Safety and efficacy of sugammadex for the reversal of rocuronium-induced neuromuscular blockade in cardiac patients undergoing noncardiac surgery. Eur J Anaesthesiol. 2009 Oct;26(10):874-84. doi: 10.1097/EJA.0b013e32832c605b. PMID 19455040
- [Background] Kizilay D, Dal D, Saracoglu KT, Eti Z, Gogus FY. Comparison of neostigmine and sugammadex for hemodynamic parameters in cardiac patients undergoing noncardiac surgery. J Clin Anesth. 2016 Feb;28:30-5. doi: 10.1016/j.jclinane.2015.08.002. Epub 2015 Nov 11. PMID 26796612
- [Result] Staikou C, Stamelos M, Stavroulakis E. Impact of anaesthetic drugs and adjuvants on ECG markers of torsadogenicity. Br J Anaesth. 2014 Feb;112(2):217-30. doi: 10.1093/bja/aet412. Epub 2013 Dec 3. PMID 24305646
- [Result] Carron M, Zarantonello F, Tellaroli P, Ori C. Efficacy and safety of sugammadex compared to neostigmine for reversal of neuromuscular blockade: a meta-analysis of randomized controlled trials. J Clin Anesth. 2016 Dec;35:1-12. doi: 10.1016/j.jclinane.2016.06.018. Epub 2016 Aug 4. PMID 27871504
- [Result] Hristovska AM, Duch P, Allingstrup M, Afshari A. The comparative efficacy and safety of sugammadex and neostigmine in reversing neuromuscular blockade in adults. A Cochrane systematic review with meta-analysis and trial sequential analysis. Anaesthesia. 2018 May;73(5):631-641. doi: 10.1111/anae.14160. Epub 2017 Dec 27. PMID 29280475
- [Result] Yamashita Y, Takasusuki T, Kimura Y, Komatsuzaki M, Yamaguchi S. Effects of Neostigmine and Sugammadex for Reversal of Neuromuscular Blockade on QT Dispersion Under Propofol Anesthesia: A Randomized Controlled Trial. Cardiol Ther. 2018 Dec;7(2):163-172. doi: 10.1007/s40119-018-0119-9. Epub 2018 Sep 14. PMID 30218410
- See also: Sugammadex briefing document — https://www.fdanews.com/ext/resources/files/11-15/110615-merck.pdf?1515434323